CLINICAL TRIAL: NCT03585582
Title: Pediatric Acute Respiratory Distress Syndrome: Determining Post-discharge Outcomes, the Effect of Early Diagnosis, and Identifying Inflammatory Signatures to Better Understand Disease Mechanism
Brief Title: Post-discharge Outcomes of Pediatric Acute Respiratory Distress Syndrome
Acronym: PARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sze Man Tse, Pediatric Respirologist, Assistant Clinical Professor, St. Justine's Hospital
Other Study IDs: MRC-155352
Record Dates: First submitted 2018-05-10; First posted 2018-07-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome
Keywords: Respiratory Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine, and tracheal or nasopharyngeal aspirate samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PARDS survivors: 1. Children <18 years
  2. diagnosed with PARDS, as defined by PALICC
  3. admitted to the ICU at the CHUSJ, a pediatric tertiary care center
  Interventions: Other: Prospective follow-up

INTERVENTIONS:
Other: Prospective follow-up — This is a prospective follow-up study to assess of outcomes at 1 year following the discharge from the hospitalization during which PARDS was diagnosed

SUMMARY:
In this study, the investigators aim to better characterize the outcomes of pediatric acute respiratory distress syndrome (PARDS) survivors, to examine whether subgroups of children with PARDS can be identified, and to determine whether an earlier diagnosis of PARDS using a computerized decision support system will improve the care of these children.

DETAILED DESCRIPTION:
Pediatric acute respiratory distress syndrome (PARDS), a heterogeneous clinical syndrome characterized by acute lung injury and hypoxemia, affects up to 10% of pediatric intensive care unit (ICU) patients and has a mortality rate of 18-27%. Because children who survived PARDS are still developing, long-term morbidities are highly relevant, although data on the outcomes of PARDS survivors is lacking. Previous studies were limited by their sample size, were outdated in PARDS management strategies, and used the adult ARDS diagnostic criteria. Some studies focused on pulmonary function but not on other patient-oriented outcomes such as respiratory symptoms, mental health issues, quality of life, and health care resource use, all of which have been identified as prevalent issues in adult ARDS survivors. Recently, adult studies have identified 2 distinct ARDS subphenotypes with differential responses to treatment using clinical and limited biological data, providing insight on the pathophysiology of ARDS. Whether these phenotypes are present in PARDS is unknown. Furthermore, integrating newer technologies such as transcriptomics in the identification of subphenotypes may improve our understanding of disease mechanisms. Finally, delays in ARDS diagnosis are common and compliance with current ARDS ventilation management guidelines is poor, ranging from 20-39% even in patients selected for clinical trials. Thus, novel methods such as decision support systems may play a role in the diagnosis and management of PARDS patients, although this remains to be evaluated.

ELIGIBILITY:
Inclusion criteria:

* clinical diagnosis of PARDS, as defined by PALICC
* aged less than 18 years
* admitted to the intensive care unit

Exclusion Criteria

- none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to the ICU at the CHUSJ, a pediatric tertiary care center
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of respiratory symptoms | At 1 year following the discharge
  Prevalence of respiratory symptoms (cough, exercise intolerance, wheezing, etc.)

SECONDARY OUTCOMES:
non-respiratory PELOD-2 score | At 7 days
  PELOD-2 score - validated score predictive of mortality (quantifies the severity of organ dysfunction). There are 7 items describing 4 organ dysfunction (respiratory component is removed). The score ranges from 0 to 25, with higher score indicating more organ dysfunction.
Pulmonary function - Forced expiratory volume in 1 second | At 1 year following the discharge
  Forced expiratory volume in 1 second (FEV1) in L and z-score based on references from the Global Lung Initiative.
Pulmonary function - Forced vital capacity (FVC) | At 1 year following the discharge
  Forced vital capacity (FVC) in L and z-score based on references from the Global Lung Initiative.
Pulmonary function - FEV1/FVC | At 1 year following the discharge
  FEV1/FVC ratio z-score based on references from the Global Lung Initiative
Pulmonary function - lung volumes | At 1 year following the discharge
  Lung volumes (total lung capacity, functional residual capacity, residual volumes) in L. Outcome measured in patients 8 years and above only.
Pulmonary function - diffusion capacity | At 1 year following the discharge
  Diffusion capacity of CO (DLCO). Outcome measured in patients 8 years and above only.
Pulmonary function - maximal inspiratory and expiratory pressures | At 1 year following the discharge
  Maximal inspiratory and expiratory pressures in cm H2O. Outcome measured in patients 6 years and above only.
Pulmonary function - resistance at 5Hz | At 1 year following the discharge
  Respiratory resistance measured using oscillometry at 5 Hz. Outcome measured in patients 3-5 years old and those who cannot perform spirometry.
Cardiopulmonary exercise testing - VO2max | At 1 year following the discharge
  VO2max measured using a standardized maximal incremental cycle ergometry protocol in children ≥ 8 years.
Cardiopulmonary exercise testing - CO2 output | At 1 year following the discharge
  CO2 output measured using a standardized maximal incremental cycle ergometry protocol in children ≥ 8 years.
Cardiopulmonary exercise testing - respiratory exchange ratio | At 1 year following the discharge
  Respiratory exchange ratio measured using a standardized maximal incremental cycle ergometry protocol in children ≥ 8 years.
Cardiopulmonary exercise testing - anaerobic threshold | At 1 year following the discharge
  Anaerobic threshold measured using a standardized maximal incremental cycle ergometry protocol in children ≥ 8 years.
Health-related quality of life - Infant Toddler Quality of Life Questionnaire | At 1 year following the discharge
  Health-related quality of life using the Infant Toddler Quality of Life Questionnaire (ages 2 months to 2 years). There are 8 scales to this 47-item questionnaire: overall health, physical abilities, growth and development, bodily pain/discomfort, temperament and mood, combined behavior, general health perceptions, change in health. There are also 3 scales that assess the impact on the parent: parental impact-emotional, parental impact-time, family cohesion. Transformed scores for all scales range from 0 to 100, with a higher score indicating better health.
Health-related quality of life - Pediatric Quality of Life Inventory | At 1 year following the discharge
  Health-related quality of life using the Pediatric Quality of Life Inventory (≥2 years), Generic core scale. There are separate versions for 2-4 year-olds (parent report only), 5-7 (parent and child report), 8-12 (parent and child report), 13-18 (parent and child report). Scores are transformed on a scale from 0 to 100, with a higher score indicating better health-related quality of life.
Mental health - Child Behavior Checklist | At 1 year following the discharge
  Mental health assessed by the parent-completed Child Behavior Checklist (age ≥ 18 months). The 6 scales are based on the DSM5: depressive problems, anxiety problems, somatic problems, attention deficit/hyperactivity problems, oppositional defiant problems, conduct problems. The raw scores are transformed into percentiles for each scale. The higher the percentile, the more problems there are.
Post-traumatic stress syndrome - Children's Impact of Event Scales | At 1 year following the discharge
  Post-traumatic stress syndrome symptoms using the Children's Impact of Event Scales (≥ 7 years). There are 8 items that are scored on a four point scale (total score from 0 to 40). A total score of 17 or more indicates symptoms suggestive of PTSD.
Post-traumatic stress syndrome - parents PTSD Checklist | At 1 year following the discharge
  Post-traumatic stress syndrome symptoms in the parents using the parents PTSD Checklist. There are 20 items that are scored from 0-4 each (total score from 0 to 80). A PCL-5 score of 33 or more indicates symptoms suggestive of PTSD.
Health resources use | At 1 year following the discharge
  Health resources use, including all-cause emergency department visits or re-hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Sze Man Tse, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- Sainte-Justine University Hospital Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No